CLINICAL TRIAL: NCT03809351
Title: UAB Alzheimer's Disease Center Core Cohort - Tau Imaging Substudy
Acronym: AV1451 ADC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jonathan E McConathy, Director, Division of Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R19-006; 1P30AG086401-01 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [F-18]AV-1451-PET/MRI (Experimental): All participants in this study will undergo a tau-PET imaging using the tracer [F-18]AV-1451 with a simultaneous PET/MRI system. The [F-18]AV-1451 dosage is 740MBq (10 mCi) given intravenously, and the PET/MRI imaging will occur 75-105 min after tracer injection.
  Interventions: Drug: [F-18]AV-1451-PET

INTERVENTIONS:
Drug: [F-18]AV-1451-PET — All study participants will undergo brain imaging with [F-18]AV-1451-PET/MRI. [F-18]AV-1451 is a PET imaging agent used primarily to measure the amount of abnormal tau protein deposition the brain.

SUMMARY:
The primary objective of this study is to measure the concentration and the regional brain distribution of pathologic tau deposition using the PET tracer AV-1451 in participants in the UAB-ADC cohort. The amount and distribution of AV-1451 in the brain will be correlated to demographic, clinical, genetic, and biospecimen data acquired through the separate ongoing UAB-ADC study. Assessment of interactions between race and vascular risk factors, brain tau levels measured with AV-1451-PET, and cognitive status will be the primary outcome of this imaging study. Individuals participating in this AV-1451-PET/MRI study will also be enrolled in an ongoing [C-11]PiB-PET/MRI study (IRB-300001005, IND-138128), and their amyloid, tau and cognitive statuses will be compared in terms of race and vascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in the UAB-ADC study under a separate IRB-approved research protocol.
2. Enrollment in the UAB-ADC amyloid-PET substudy under a separate IRB-approved research protocol. The amyloid-PET study does not have to have been completed prior to enrollment and participation in this tau-PET study.
3. Negative urine or serum hCG test within 2 days of [F-18]AV-1451 administration in women of child bearing potential. Women who are post-menopausal with at least 1 year since last menses or documented surgical sterilization will not require pregnancy testing.

Exclusion Criteria:

1. Meets any exclusion criteria for the UAB-ADC study.
2. Inability or contraindication for undergoing MRI and/or PET imaging
3. Inability to participate in the imaging studies due to severity of dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of pathological tau deposition in the brain. | 5 years
  The amount and regional distribution of pathological tau in the brains of study participants will be measured with [F-18]AV-1451-PET/MRI using standardized uptake value ratios (SUVRs) derived from the PET images.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States